CLINICAL TRIAL: NCT06687967
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Investigate the Efficacy and Safety of Dupilumab for the Treatment of Pruritus of Lichen Simplex Chronicus (LSC) in Adults
Brief Title: A Study to Investigate Improvement in Pruritus of Lichen Simplex Chronicus With Dupilumab Injections Compared With Placebo in Male and Female Participants Aged at Least 18 Years (STYLE 1)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC18365; 2024-514737-37-00 (Registry Identifier: CTIS); U1111-1307-7329 (Registry Identifier: WHO ICTRP)
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lichen Simplex Chronicus
MeSH Terms: conditions — Neurodermatitis | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dupilumab (Experimental): Dupilumab subcutaneous injection as per protocol
  Interventions: Drug: Dupilumab
- Placebo (Placebo Comparator): Placebo subcutaneous injection as per protocol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab — Pharmaceutical form: Solution for injection Route of administration: subcutaneous injection
  Other Names: SAR231893; Dupixent
  Arms: Dupilumab
Drug: Placebo — Pharmaceutical form: Solution for injection Route of administration: subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a parallel, Phase 3, 2-arm study for treatment. The purpose of this study is to measure improvement in pruritus with dupilumab subcutaneous injections compared with placebo injections in male and female participants aged at least 18 years with LSC.

Study details include:

The study duration will be up to 40 weeks. The treatment duration will be up to 24 weeks. The follow-up duration after treatment will be 12 weeks. The number of visits will be 6.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply (at screening and baseline unless otherwise specified):

* Participant must be at least 18 years of age or the legal age of consent in the jurisdiction in which the study is taking place at the time of signing the informed consent.
* Participants with moderate-to-severe LSC, as defined by Investigator's Global Assessment (IGA) score ≥3 and one or more of the following:

  * at least 1 single anogenital lesion;
  * at least 2 lesions including 1 lesion of ≥3 cm in diameter;
  * at least 1 severe lesion (IGA score = 4).
* History of LSC for at least 6 months prior to the screening visit.
* On the Worst-Itch Numerical Rating Scale (WI-NRS) ranging from 0 to 10, participants must have an average worst-itch of LSC score of ≥7 in the 7 days prior to Day 1. A minimum of 4 daily scores out of the 7 days is required to calculate the baseline average score. For participants who do not have at least 4 daily scores reported during the 7 days immediately preceding the planned randomization date, randomization can be postponed until this requirement is met, but without exceeding the 28-day maximum duration of the screening period.
* History of failing a 2-week course of medium-to-superpotent topical corticosteroid (TCS) +/- topical calcineurin inhibitor (TCI) for the treatment of LSC within the last 6 months, unless TCS/TCI are medically not advisable. Patients with documented systemic treatment for LSC (other than antihistamines) in the past 6 months are also considered as inadequate responders to topical treatments and are potentially eligible for treatment with dupilumab after appropriate washout.
* Appropriate contraceptive measures

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply (at screening and baseline unless otherwise specified):

* Participants diagnosed with active lesions of prurigo nodularis (broadly distributed nodules) or active lesions of atopic dermatitis (AD) within 6 months, contact dermatitis, psoriasis, cutaneous T-cell lymphoma (CTCL) XE "CTCL" \f Abbreviation \t "cutaneous T-cell lymphoma" (or suspected of CTCL), vulvar lichen planus, or vulvar lichen sclerosus.
* Presence of skin morbidities other than LSC that, in the opinion of the Investigator, may interfere with the assessment of the study outcomes. For example: scabies, insect bite, folliculitis, lymphomatoid papulosis, chronic actinic dermatitis, dermatitis herpetiformis, sporotrichosis, bullous disease, lichen planus hypertrophicus.
* Severe concomitant illness(es) that, in the Investigator's judgment, would adversely affect the participant's participation in the study.
* Severe psychiatric disease that, in the Investigator's judgement, would affect the study intervention evaluation.
* Having received or planning to use any of the treatments within the timeframe as specified in the protocol.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2024-11-28 (Actual); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with improvement (reduction) in weekly average of daily WI-NRS by ≥4 from baseline to Week 24 | Week 24
  Worst-Itch numerical rating score (WI-NRS) is a patient report outcome (PRO) comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").

SECONDARY OUTCOMES:
Absolute change in weekly average of daily WI-NRS from baseline to Week 24 | Baseline to Week 24
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Percentage change in weekly average of daily WI-NRS from baseline to Week 24 | Baseline to Week 24
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Absolute change in weekly average of daily Itch-related Sleep Disturbance NRS from baseline to Week 24 | Baseline to Week 24
  The Itch-related Sleep Disturbance NRS is a single-item PRO to report the degree of sleep loss related to itch over the past 24 hours, from 0 ("no sleep loss related to itch") to 10 ("I cannot sleep at all due to itch").
Percentage change in weekly average of daily Itch-related Sleep Disturbance NRS from baseline to Week 24 | Baseline to Week 24
  The Itch-related Sleep Disturbance NRS is a single-item PRO to report the degree of sleep loss related to itch over the past 24 hours, from 0 ("no sleep loss related to itch") to 10 ("I cannot sleep at all due to itch").
Absolute change in ItchyQoL score from baseline to Week 24 | Baseline to Week 24
  Itchy quality of life survey (ItchyQoL) is a pruritus-specific QoL instrument to measure dermatology-specific QoL in patients aged 16 years and older. The overall score ranging from 1 to 5. A higher score corresponds to a more adverse impact on health-related QoL
Absolute change in DLQI total score from baseline to Week 24 | Baseline to Week 24
  Dermatology life quality index (DLQI) is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer health-related QoL.
Proportion of participants with improvement (reduction) in weekly average of daily WI-NRS by ≥4 from baseline to Week 12 | Week 12
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Proportion of participants with IGA 0 or 1 score for LSC at Week 12 and Week 24 | Week 12 and 24
  Investigator's Global Assessment (IGA) for LSC is a clinician-reported outcome using a 5-point scale from 0 (clear) to 4 (severe)
Proportion of participants with both an improvement (reduction) in weekly average of daily WI-NRS by ≥4 from baseline to Week 24 and an IGA 0 or 1 score for LSC at Week 24 | Baseline through Week 24
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch"). IGA for LSC is a clinician-reported outcome using a 5-point scale from 0 (clear) to 4 (severe).
Incidence of treatment-emergent anti-drug antibody (ADA) against dupilumab | Baseline through Week 36
Percentage of participants experiencing treatment-emergent adverse event (TEAEs) or serious adverse event (SAEs) | Baseline through Week 36

CONTACTS AND LOCATIONS:
Locations (63):
- United States (11):
  - Dermatology Research Associates - Los Angeles- Site Number : 8400004, Los Angeles, California
  - Quality Care Clinical Research- Site Number : 8400034, Miami, Florida
  - Michigan Center for Research Company- Site Number : 8400013, Clarkston, Michigan
  - JDR Dermatology Research- Site Number : 8400023, Las Vegas, Nevada
  - Equity Medical- Site Number : 8400017, New York, New York
  - Onsite Clinical Solutions - Huntersville- Site Number : 8400033, Huntersville, North Carolina
  - Wake Forest University Health Sciences- Site Number : 8400028, Winston-Salem, North Carolina
  - Red River Research Partners - Fargo- Site Number : 8400007, Fargo, North Dakota
  - Center for Clinical Studies - Houston - Binz Street- Site Number : 8400011, Houston, Texas
  - MedCare Pharma - Houston - Cypress Creek Parkway- Site Number : 8400014, Houston, Texas
  - Care Access - Arlington- Site Number : 8400022, Arlington, Virginia
- Argentina (4):
  - Investigational Site Number : 0320003, Rosario, Santa Fe Province
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320002, Mendoza
- Canada (7):
  - Investigational Site Number : 1240005, Edmonton, Alberta
  - Investigational Site Number : 1240001, London, Ontario
  - Investigational Site Number : 1240007, Mississauga, Ontario
  - Investigational Site Number : 1240009, Montreal, Quebec
  - Investigational Site Number : 1240008, Québec, Quebec
  - Investigational Site Number : 1240010, Regina, Saskatchewan
  - Investigational Site Number : 1240002, Saskatoon, Saskatchewan
- Chile (3):
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
- China (5):
  - Investigational Site Number : 1560002, Beijing
  - Investigational Site Number : 1560004, Hangzhou
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560003, Shijiazhuang
  - Investigational Site Number : 1560005, Suzhou
- Investigational Site Number : 2030001, Ostrava, Czechia
- Germany (2):
  - Investigational Site Number : 2760003, Bad Bentheim
  - Investigational Site Number : 2760001, Magdeburg
- Greece (3):
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000002, Thessaloniki
  - Investigational Site Number : 3000003, Thessaloniki
- Hungary (2):
  - Investigational Site Number : 3480001, Debrecen
  - Investigational Site Number : 3480002, Kaposvár
- Italy (2):
  - Investigational Site Number : 3800001, Rome, Roma
  - Investigational Site Number : 3800002, Bologna
- Japan (6):
  - Investigational Site Number : 3920002, Ebina-shi, Kanagawa
  - Investigational Site Number : 3920001, Kamiamakusa, Kumamoto
  - Investigational Site Number : 3920007, Sakai, Osaka
  - Investigational Site Number : 3920003, Tachikawa, Tokyo
  - Investigational Site Number : 3920009, Fukuoka
  - Investigational Site Number : 3920005, Kagoshima
- Mexico (2):
  - Investigational Site Number : 4840003, Aguascalientes
  - Investigational Site Number : 4840001, Chihuahua City
- Portugal (3):
  - Investigational Site Number : 6200002, Coimbra
  - Investigational Site Number : 6200003, Lisbon
  - Investigational Site Number : 6200001, Porto
- Spain (4):
  - Investigational Site Number : 7240003, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240005, Barcelona, Catalunya [Cataluña]
  - Investigational Site Number : 7240002, Barcelona, Catalunya [Cataluña]
  - Investigational Site Number : 7240004, Valencia
- Taiwan (3):
  - Investigational Site Number : 1580002, Kaohsiung City
  - Investigational Site Number : 1580003, New Taipei City
  - Investigational Site Number : 1580001, Taipei
- Turkey (Türkiye) (3):
  - Investigational Site Number : 7920003, Adapazarı
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920001, Samsun
- United Kingdom (2):
  - Investigational Site Number : 8260002, Milton Keynes, Buckinghamshire
  - Investigational Site Number : 8260001, London, England

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC18365 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26222&tenant=MT_SNY_9011